CLINICAL TRIAL: NCT02252718
Title: Amsterdam Stool Scale: Usefulness in Clinical Setting
Status: Completed | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Katarzyna Wojtyniak, M.D., Medical University of Warsaw
Other Study IDs: 1-2014
Record Dates: First submitted 2014-09-23; First posted 2014-09-30 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Stool Assessment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children 1-18 months of age: Children aged between 1 month and 18 months admitted to the Department of Pediatrics The Medical University of Warsaw
  Interventions: Other: Stool Assessment

INTERVENTIONS:
Other: Stool Assessment — After passing a stool by the child participating in the study, within a short-time interval (<5 min), the stool will be assessed independently by one of the parents and the medical doctor. At the same time a parent will take 2 photos with phone photographic camera. Then the photographs will be independently evaluated by another doctor who will be unaware of both the "in vivo" stool appraisal and child condition.

SUMMARY:
The aim of this study is to assess interobserver and intraobserver variability of the Amsterdam Stool Scale in clinical practice. After passing a stool by the child participating in the study it will be assessed using the Amsterdam Stool Scale independently by one of the parents and the medical doctor. At the same time a parent will take 2 photos that will be independently evaluated by another doctor.

DETAILED DESCRIPTION:
INTRODUCTION:

Description of stool appearance is important in clinical practice. Parents are often asked to evaluate stool of their child. At present parents also take more frequently photos using smartphone camera when they are concerned with child's stool appearance and show it to their doctors. To make stool evaluation easier there have been stool form scales created. One of this is Amsterdam Stool Scale that enables stool assessment of children who are not yet toilet trained. This scale facilitates to describe amount, consistency and color of the stool.

AIM:

To assess interobserver and intraobserver variability of the Amsterdam Stool Scale in clinical practice.

METHODS:

After passing a stool by the child participating in the study, within a short-time interval (<5 min), the stool will be assessed independently by one of the parents and the medical doctor. At the same time a parent will take 2 photos with phone camera. The photographs then will be independently evaluated by another doctor who will be unaware of both the "in vivo" stool appraisal and child condition.

STATISTICAL ANALYSIS:

Then the interobserver (between a parent, the doctor and the doctor assessing photograph) variability will be evaluated by calculating the kappa (κ) statistics for nominal data for the stool consistency, amount and color separately.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-18 months of age
* Lack of ability to use the toilet

Exclusion Criteria:

* Lack of parental consent to participate in the study
* Parental inability to understand the study procedures

Ages: 1 Month to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The group will be selected from the children admitted to the Department of Pediatrics The Medical University of Warsaw
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Paediatrics, The Medical University of Warsaw, Warsaw, Poland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at the Department of Paediatrics of the Medical University of Warsaw between September 2014 and February 2015.
Groups:
- Children 2-18 Months of Age: Children aged between 2 and 18 months of age, who were not toilet trained, admitted to the Department of Pediatrics The Medical University of Warsaw
  Stool Assessment: After passing a stool by the child participating in the study, within the shortest possible time (<5 min), the stool will be assessed independently and simulataneously by one of the parents and the medical doctor. They were unaware of the evaluation results made by the other. At the same time 2 photos were taken with smartphone camera. Then the photographs were subsequently evaluated by the other physician (MD2), who was unaware of the in vivo stool evaluation.
Period: Overall Study
Arm/Group | Children 2-18 Months of Age
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Children between 2 and 18 months of age who were not toilet trained were eligible for the study. Exclusion criteria included parental inability to understand the study procedure and lack of parental consent to participate.
Groups:
- Children 2-18 Months of Age: Children between 2 and 18 months of age who were not toilet trained
Arm/Group | Children 2-18 Months of Age
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: month] | 5.02 (4.4)
Gender [Count of Participants; unit: Participants]
  Female | 42
  Male | 58

OUTCOME MEASURES:

1. Primary Outcome: Interrater Variability (IV)
Description: The outcome measures were interrater variability in the stool assessment by the parent and MD1 made in vivo and in the assessment by the parent in vivo and by MD2 based on the photograph(s). The IV was evaluated by calculating the proportion of exact agreement and the κ statistics for nominal data (colour) and weighted κ values for items in which there is a natural ordering of categories (consistency and amount). Correlation, based on the value of kappa (κ), was categorized as poor (κ ≤ 0.2), fair (0.21 ≤ κ ≤ 0.40), moderate (0.41 ≤ κ ≤ 0.60), good (0.61 ≤ κ ≤ 0.80) or excellent (0.81 ≤ κ ≤ 1.00).
Time Frame: <5min after defecation
Measure: Number (95% Confidence Interval); unit: kappa value
Arm/Group | Children 2-18 Months of Age
Number analyzed (Participants) | 100
kappa value
  parent- MD1: amount | 0.79 [0.7 to 0.88]
  parent- MD1: consistency | 0.87 [0.78 to 0.95]
  parent- MD1: color | 0.81 [0.71 to 0.91]
  parent- MD2: amount | 0.44 [0.3 to 0.59]
  parent- MD2: consistency | 0.5 [0.36 to 0.64]
  parent- MD2: color | 0.33 [0.21 to 0.45]

ADVERSE EVENTS:
Arm/Group | Children 2-18 Months of Age
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 0/100

LIMITATIONS AND CAVEATS:
Limitations of our study included the lack of external validity. Children were recruited in only one paediatric department. Only one physician conducted stool assessment in vivo and only one physician evaluated photographs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes